CLINICAL TRIAL: NCT01605825
Title: A Phase 2b Study of Dalfampridine 10mg Extended Release Tablet in Subjects With Chronic Deficits After Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DALF-PS-1003
Record Dates: First submitted 2012-05-21; First posted 2012-05-25 (Estimated); Results first posted 2014-03-10 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2015-12

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- placebo/dalfampridine-ER (Placebo Comparator): Subjects will be randomized at day 1 to one of two blinded treatment sequences (A or B) in a 2:1 ratio respectively, according to a randomization created prior to the start of the study:
  Period 1 = days 1, 8 and 15. Period 2 = Days 22, 29, and 36
  Interventions: Drug: placebo/dalfampridine-ER
- dalfampridine-ER/placebo (Placebo Comparator): Subjects will be randomized at day 1 to one of two blinded treatment sequences (A or B) in a 2:1 ratio respectively, according to a randomization created prior to the start of the study:
  Period 1 = days 1, 8 and 15. Period 2 = Days 22, 29, and 36
  Interventions: Drug: dalfampridine-ER/placebo

INTERVENTIONS:
Drug: placebo/dalfampridine-ER — Sequence A: placebo in Period 1 and dalfampridine-ER in Period 2. 10mg tablets, will be taken orally, twice daily approximately 12 hours apart
  Arms: placebo/dalfampridine-ER
Drug: dalfampridine-ER/placebo — Sequence B: dalfampridine-ER in Period 1 and placebo in Period 2. 10mg tablets, will be taken orally, twice daily approximately 12 hours apart
  Arms: dalfampridine-ER/placebo

SUMMARY:
This is a multi-center, safety and tolerability study in subjects with chronic stable sensorimotor deficits after ischemic stroke. It has been designed as a double-blind, placebo-controlled, 2-period crossover study.

ELIGIBILITY:
Inclusion Criteria:

* History of a stable sensorimotor deficit due to an ischemic stroke, as confirmed by the Investigator with supportive prior imaging findings (MRI/ CT scan)
* ≥ 6 months post-stroke
* Have a body mass index (BMI) ranging between 18.0 - 35.0 kg/m,2 inclusive
* Stable concomitant medication therapy regimen within 4 weeks of screening visit

Exclusion Criteria:

* History of seizures, except simple febrile seizures
* Moderate or severe renal impairment as defined by a calculated creatinine clearance of ≤ 50 mL/minute using the Cockcroft-Gault Equation
* Botulinum toxin use within 2 months prior to the Screening Visit
* Orthopedic surgical procedures in any of the extremities within the past 6 months
* Diagnosis of multiple sclerosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2012-05; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathews Adera, MD, Study Director — Acorda Therapeutics
Locations (20):
- United States (20):
  - Acorda Site #011, Birmingham, Alabama
  - Acorda Site #018, La Jolla, California
  - Acorda Site #016, Newport Beach, California
  - Acorda Site #006, Fairfield, Connecticut
  - Acorda Site #002, Atlantis, Florida
  - Acorda Site #015, Fort Lauderdale, Florida
  - Acorda Site #003, Decatur, Georgia
  - Acorda Site #021, Lexington, Kentucky
  - Acorda Site #009, Boston, Massachusetts
  - Acorda Site #017, Saginaw, Michigan
  - Acorda Site #020, Great Falls, Montana
  - Acorda Site #023, Reno, Nevada
  - Acorda Site #022, New Brunswick, New Jersey
  - Acorda Site #019, Buffalo, New York
  - Acorda Site #007, West Haverstraw, New York
  - Acorda Site #004, White Plains, New York
  - Acorda Site #013, Charlotte, North Carolina
  - Acorda Site #001, Philadelphia, Pennsylvania
  - Acorda Site #008, Norfolk, Virginia
  - Acorda Site #010, Bellevue, Washington

REFERENCES:
- [Derived] Iaci JF, Parry TJ, Huang Z, Finklestein SP, Ren J, Barrile DK, Davenport MD, Wu R, Blight AR, Caggiano AO. Dalfampridine improves sensorimotor function in rats with chronic deficits after middle cerebral artery occlusion. Stroke. 2013 Jul;44(7):1942-50. doi: 10.1161/STROKEAHA.111.000147. Epub 2013 May 7. PMID 23652269

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo/Dalfampridine-ER: Subjects will be randomized at day 1 to one of two blinded treatment sequences (A or B) in a 2:1 ratio respectively, according to a randomization created prior to the start of the study:
  Period 1 = days 1, 8 and 15. Period 2 = Days 22, 29, and 36
  dalfampridine-ER: Sequence A: placebo in Period 1 and dalfampridine-ER in Period 2.
  10mg tablets, will be taken orally, twice daily approximately 12 hours apart
- Dalfampridine-ER/Placebo: Subjects will be randomized at day 1 to one of two blinded treatment sequences (A or B) in a 2:1 ratio respectively, according to a randomization created prior to the start of the study:
  Period 1 = days 1, 8 and 15. Period 2 = Days 22, 29, and 36
  dalfampridine-ER: Sequence B: dalfampridine-ER in Period 1 and placebo in Period 2.
  10mg tablets, will be taken orally, twice daily approximately 12 hours apart
Period: Overall Study
Arm/Group | Placebo/Dalfampridine-ER | Dalfampridine-ER/Placebo
Started | 55 | 28
Completed | 45 | 25
Not Completed | 10 | 3
Not completed — Adverse Event | 4 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Non-Compliance -Investigational Drug | 3 | 0
Not completed — Non-Compliance with Protocol | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: The Safety Population consists of all randomized subjects who took at least one dose of investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo/Dalfampridine-ER | Dalfampridine-ER/Placebo | Total
Number analyzed (Participants) | 55 | 28 | 83
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (9.72) | 63.5 (8.91) | 59.5 (9.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 10 | 28
  Male | 37 | 18 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 15 | 4 | 19
  White | 38 | 22 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Dalfampridine-ER in Subjects With Chronic Deficits After Ischemic Stroke Assessed by Number of Treatment Emergent Adverse Events (TEAEs)
Description: A TEAE is defined as any adverse event with date of onset (or worsening) on or after the start-date of double-blind treatment through 7 days after the last dose of double-blind treatment.
  The severity categories of mild, moderate or severe, are defined below:
  * Mild is defined as causing no limitation of usual activities
  * Moderate is defined as causing some limitation of usual activities
  * Severe is defined as causing inability to carry out usual activities
Time Frame: up to 36 days
Population: Safety population. Number of participants analyzed is number of patients with TEAE's as described in outcome measure description. Excludes pre-treatment and post-treatment adverse events.
Measure: Number; unit: participants
Arm/Group | Placebo | Dalfampridine-ER
Number analyzed (Participants) | 81 | 77
participants
  Subjects with any TEAEs | 30 | 42
  TEAEs Possibly Related to study drug | 16 | 24
  TEAEs Maximum Severity - Mild | 16 | 29
  TEAEs Maximum Severity - Moderate | 13 | 10
  TEAEs Maximum Severity - Severe | 1 | 3
  TEAEs leading to withdrawal of study drug | 1 | 5
  TEAEs Serious | 2 | 2
  Subjects who died | 0 | 0

2. Other Pre Specified Outcome: Walking Speed Measured by the Timed 25 Foot Walk Test (T25FW)
Time Frame: Screening visit, Days 1, 8, 15, 22, 29 and 36
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Motor and Sensory Function as Measured by the Fugl-Meyer Assessment (FMA)
Time Frame: Screening visit, Days 1, 8, 15, 22, 29, and 36
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Manual Dexterity as Measured by the Box and Block Test
Time Frame: Days 1, 8, 15, 22, 29, and 36
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Assistance Required to Perform Activities of Daily Living (ADL) by the Functional Independence Measure (FIM) Scale
Time Frame: Days 1, 8, 15, 22, 29, and 36
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Subject Global Impression (SGI) Scale
Time Frame: Days 8, 15, 22, 29 and 36
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Clinician Global Impression (CGI) Scale
Time Frame: Days 8, 15, 22, 29 and 36
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Hand Strength as Measured by the Grip Test and Pinch Tests
Time Frame: Days 1, 8, 15, 22, 29, and 36
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: up to 36 days
Description: All adverse events discussed in this report are treatment-emergent adverse events (TEAEs) unless otherwise indicated. Therefore, events that had a date of onset, or worsening, on or after start of double-blind treatment through 7 days after the last dose of double-blind treatment
Arm/Group | Placebo | Dalfampridine-ER
Serious Adverse Events (participants affected / at risk) | 2/81 | 2/77
Other Adverse Events (participants affected / at risk) | 30/81 | 42/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Dalfampridine-ER (N=77)
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 2
Suicide attempt (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=81) | Dalfampridine-ER (N=77)
Dizziness (Nervous system disorders) | 2 | 8
Nausea (Gastrointestinal disorders) | 5 | 3
Fatigue (General disorders) | 3 | 4
Insomnia (Psychiatric disorders) | 2 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Asthenia (General disorders) | 1 | 3
Constipation (Gastrointestinal disorders) | 4 | 0
Headache (Nervous system disorders) | 3 | 2
Convulsion (Nervous system disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Drooling (Nervous system disorders) | 3 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Chest pain (General disorders) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Depression (Psychiatric disorders) | 2 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 2
Gait disturbance (General disorders) | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pain (General disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Tremor (Nervous system disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has the right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.